CLINICAL TRIAL: NCT02554773
Title: An Open-label Extension Study of Subcutaneously Administered Fitusiran in Patients With Moderate or Severe Hemophilia A or B Who Have Participated in a Previous Clinical Study With Fitusiran
Brief Title: An Open-label Extension Study of an Investigational Drug, Fitusiran, in Patients With Moderate or Severe Hemophilia A or B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTE14762; ALN-AT3SC-002 (Other: Alnylam); 2015-001395-21 (EudraCT Number); U1111-1251-5204 (Registry Identifier: ICTRP)
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; RNAi therapeutic
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fitusiran (Experimental): Patients will be administered subcutaneous (SC) fitusiran once monthly or every 2 months according to the dose selection rules defined in protocol.
  Interventions: Drug: Fitusiran (SAR439774)

INTERVENTIONS:
Drug: Fitusiran (SAR439774) — Pharmaceutical form: solution for injection Route of administration : subcutaneous (sc)

SUMMARY:
Primary Objective:

To evaluate the long-term safety and tolerability of fitusiran in male patients with moderate or severe hemophilia A or B

Secondary Objectives:

* To investigate the long-term efficacy of fitusiran
* To characterize the safety and efficacy of concomitantly administered Factor VIII (FVIII), Factor IX (FIX) or bypassing agents (BPA) and fitusiran for treatment of bleeding episodes
* To assess changes in health-related quality of life (QOL) over time
* To characterize antithrombin (AT) reduction and thrombin generation (TG) increase
* To characterize the pharmacokinetics (PK) of fitusiran

DETAILED DESCRIPTION:
It is anticipated that patients in this study will receive treatment with open label fitusiran for approximately 7 years or until fitusiran becomes commercially available, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Completed and tolerated study drug dosing in study TDR14767 (ALN-AT3SC-001)
* Male aged ≥18 years
* Moderate or severe, clinically stable hemophilia A or B as evidenced by a laboratory FVIII or FIX level ≤5% at screening. Patients with a FVIII or FIX level >5% at screening will be eligible on provision of a historic laboratory report indicating a trough level ≤5%
* Willing and able to comply with the study requirements and provide written informed consent

Exclusion Criteria:

* Clinically significant liver disease
* Patients known to be human immunodeficiency virus seropositive and have a CD4 count <200 cells/μL
* History of venous thromboembolism
* Current serious mental illness that, in the judgment of the Investigator, may compromise patient safety, ability to participate in all study assessments, or study integrity
* Clinically relevant history or presence of cardiovascular, respiratory, gastrointestinal, renal, neurological, inflammatory, or other diseases that, in the judgment of the Investigator, precludes study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, MD, Study Director — Sanofi
Locations (11):
- United States (2):
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Pittsburgh, Pennsylvania
- Bulgaria (2):
  - Clinical Trial Site, Plovdiv
  - Clinical Trial Site, Sofia
- Russia (2):
  - Clinical Trial Site, Kirov
  - Clinical Trial Site, Moscow
- Clinical Trial Site, Zurich, Switzerland
- United Kingdom (4):
  - Clinical Trial Site, Basingstoke
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, London
  - Clinical Trial Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pipe SW, Lissitchkov T, Georgiev P, Mangles S, Hegemann I, Trinchero A, Chowdary P, Forbes A, Feng L, Menapace LA, Kichou S, Andersson S, Demissie M, Ragni MV. Long-term safety and efficacy of fitusiran prophylaxis, and perioperative management, in people with hemophilia A or B. Blood Adv. 2025 Mar 11;9(5):1147-1158. doi: 10.1182/bloodadvances.2024013900. PMID 39642315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in 5 countries between 18 September 2015 and 21 March 2023. A total of 34 participants were enrolled in this study.
Pre-assignment Details: Participants were rolled over from the parent study TDR14767 (NCT02035605).
Groups:
- Original Dose Regimen [Safety Analysis Set 1 (SAS 1)]: Participants received fitusiran 50 milligram (mg) or 80 mg subcutaneous (SC) injection every month (QM) under the original dose and regimen.
- Antithrombin (AT)-Based Dose Regimen [Safety Analysis Set 2 (SAS 2)]: Participants received fitusiran 50 mg QM, 80 mg QM or 50 mg every 2 months (Q2M) SC injection under recommended AT-based dose regimen.
Period: Original Dose Regimen (SAS 1)
Arm/Group | Original Dose Regimen [Safety Analysis Set 1 (SAS 1)] | Antithrombin (AT)-Based Dose Regimen [Safety Analysis Set 2 (SAS 2)]
Started | 34 | 0
Completed | 18 | 0
Not Completed | 16 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Death | 1 | 0
Not completed — Other | 4 | 0
Period: AT-Based Dose Regimen (SAS 2)
Arm/Group | Original Dose Regimen [Safety Analysis Set 1 (SAS 1)] | Antithrombin (AT)-Based Dose Regimen [Safety Analysis Set 2 (SAS 2)]
Started | 0 (No participants continued to receive fitusiran under the original dose and regimen after protocol amendment 08.) | 18 (Participants who resumed fitusiran under the recommended AT-based dose regimen after protocol amendment 08.)
Completed | 0 | 12
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — More than 1 AT measurement <15% | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set 1 included all participants who received at least a partial dose of study drug during the LTE14762 study under the original dose and regimen.
Groups:
- Original Dose Regimen (SAS 1): Participants received fitusiran 50 mg or 80 mg SC injection QM under the original dose and regimen.
Arm/Group | Original Dose Regimen (SAS 1)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 33
  Asian/Oriental | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An SAE is any untoward medical occurrence that results: death or life-threatening or inpatient hospitalization or prolongation of existing hospitalization or persistent or significant disability or congenital anomaly or medically important event. All AEs collected in LTE14762 were considered TEAE because all participants received dose in the parent study. AEs of special interest (AESI) are alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations >3× upper limit of normal (ULN) or suspected or confirmed thromboembolic events or severe or serious injection site reactions or systemic injection associated reactions or cholecystitis or cholelithiasis.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: Safety analysis set (SAS) included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- AT-Based Dose Regimen (SAS 2): Participants received fitusiran 50 mg QM, 80 mg QM or 50 mg Q2M SC injection under recommended AT-based dose regimen.
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants
  Any TEAE | 33 | 14
  Any Treatment-emergent SAE | 13 | 1
  Any Treatment-emergent AESI | 11 | 1
  Any TEAE leading to study drug discontinuation | 5 | 1
  Any TEAE leading to death | 1 | 0

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality (PCSA): Hematology
Description: Blood samples were collected to determine the hematology laboratory significant abnormalities. Here, DFB = decrease from baseline, NB = non-black, and B = black.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants
  Hemoglobin: <= 115 gram per liter (g/L) | 5 | 2
  Hemoglobin: >= 185 g/L | 3 | 1
  Hemoglobin: DFB >= 20 g/L | 10 | 3
  Hematocrit: <= 0.37 fraction of 1 | 8 | 3
  Hematocrit: >= 0.55 fraction of 1 | 5 | 2
  Erythrocyte Count: >= 6 x 10^12/L | 9 | 3
  Platelet Count: < 100 x 10^9/L | 2 | 0
  Leukocyte Count: <3 x 10^9/L (NB); <2 x 10^9/L (B) | 3 | 1
  Leukocyte Count: >= 16 x 10^9/L | 1 | 1
  Neutrophils: <1.5 x 10^9/L (NB); <1 x 10^9/L (B) | 8 | 2
  Lymphocytes: > 4 x 10^9/L | 0 | 1
  Monocytes: > 0.7 x 10^9/L | 15 | 3
  Basophils: > 0.1 x 10^9/L | 4 | 0
  Eosinophils:>0.5x10^9/L or >ULN (ULN >=0.5x10^9/L) | 11 | 1

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality: Clinical Chemistry
Description: Blood samples were collected to determine the clinical chemistry laboratory abnormalities. Here, mmol/L = millimoles per liter, LLN = lower limit of normal, mg/L = milligram per liter, umol/L = micromoles per liter, mL/min = milliliter per minute, m^2 = meter square, CB = conjugated bilirubin, and DB = direct bilirubin.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants
  Glucose: <= 3.9 mmol/L and < LLN | 13 | 2
  Glucose:>=11.1 mmol/L(unfasted);>=7 mmol/L(fasted) | 10 | 2
  C-Reactive Protein: > 2 ULN or > 10 mg/L | 20 | 7
  Sodium: <= 129 mmol/L | 1 | 0
  Potassium: < 3 mmol/L | 2 | 0
  Potassium: >= 5.5 mmol/L | 5 | 0
  Creatinine: >= 150 umol/L | 1 | 1
  Creatinine: >= 30% change from baseline | 13 | 7
  Creatinine: >= 100% change from baseline | 2 | 1
  Creatinine Clearance: >= 60 - < 90 mL/min/1.73m^2 | 18 | 2
  Creatinine Clearance: >= 15 - < 30 mL/min/1.73m^2 | 1 | 1
  Uric Acid: < 120 umol/L | 2 | 0
  Uric Acid: > 408 umol/L | 20 | 8
  ALT: > 1 ULN | 30 | 6
  ALT: > 3 ULN | 14 | 1
  ALT: > 5 ULN | 6 | 1
  ALT: > 10 ULN | 2 | 0
  ALT: > 20 ULN | 1 | 0
  AST: > 1 ULN | 22 | 7
  AST: > 3 ULN | 8 | 1
  AST: > 5 ULN | 5 | 0
  AST: > 10 ULN | 1 | 0
  Alkaline Phosphatase: > 1.5 ULN | 4 | 0
  Total Bilirubin: > 1.5 ULN | 4 | 2
  CB: DB >35% Bilirubin and Bilirubin >1.5 ULN | 3 | 1

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality: Urinalysis
Description: Urine samples collected to determine the significant abnormalities in urine.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality: Vital Signs
Description: Participants vital signs were examined to determine the abnormalities. Vital signs included weight, supine systolic blood pressure (SSBP) and supine diastolic blood pressure (SDBP). Here, mmHg = millimeter of mercury, and IFB = increase from baseline.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants
  SSBP: >= 160 mmHg; IFB >= 20 mmHg | 1 | 0
  SDBP: <= 45 mmHg; DFB >= 20 mmHg | 1 | 0
  Weight: >= 5% DFB | 8 | 3
  Weight: >= 5% IFB | 15 | 9

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality: Electrocardiogram (ECG)
Description: Standard 12-lead ECGs were recorded after at least 15 minutes in the supine position using an electrocardiographic device. The following were assessed: heart rate, rhythm, interval between the peaks of successive QRS complexes (RR), interval from the beginning of the P wave until the beginning of the QRS complex (PR), interval from start of the Q wave to the end of the S wave (QRS), interval between the start of the Q wave and the end of the T wave (QT), QT interval corrected for heart rate (QTc) automatic correction evaluation, QRS axis, left ventricular hypertrophy criteria, right ventricular hypertrophy criteria, repolarization charges, and overall cardiac impression for each participant. Here, msec = milliseconds.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants
  Ventricular Rate: < 50 beats/min | 1 | 0
  Ventricular Rate: > 90 beats/min | 8 | 5
  Ventricular Rate: >90 beats/min;IFB >=20 beats/min | 3 | 1
  Ventricular Rate: > 100 beats/min | 5 | 1
  Ventricular Rate:>100 beats/min;IFB >=20 beats/min | 1 | 0
  PR Interval: > 200 msec | 3 | 0
  PR Interval: > 200 msec; IFB >= 25% | 2 | 0
  PR Interval: > 220 msec | 2 | 0
  PR Interval: > 220 msec; IFB >= 25% | 2 | 0
  PR Interval: > 240 msec | 2 | 0
  PR Interval: > 240 msec;IFB >= 25% | 2 | 0
  QRS Interval: > 110 msec | 8 | 3
  QRS Interval: > 110 msec; IFB >= 25% | 3 | 0
  QRS Interval: > 120 msec | 3 | 2
  QRS Interval: > 120 msec; IFB >= 25% | 3 | 0
  QTc Bazett: > 450 msec | 2 | 4
  QTc Bazett: > 480 msec | 1 | 1
  QTc Bazett: IFB (30-60) msec | 8 | 4
  QTc Fridericia: > 450 msec | 1 | 1
  QTc Fridericia: > 480 msec | 0 | 1
  QTc Fridericia: IFB (30-60) msec | 4 | 4

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormality: Physical Examination
Description: Physical examination included, at a minimum, an assessment of the participant's general appearance; skin; head, eyes, ears, nose, and throat; examinations of lymph nodes, abdomen, extremities/joints, neurological and mental status; heart and respiratory auscultation; peripheral arterial pulse; and pupil, knee, achilles, and plantar reflexes.
Time Frame: From first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The SAS included all participants who received at least a partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
Participants | 17 | 2

8. Secondary Outcome: Annualized Bleeding Rate (ABR) During the Efficacy Period
Description: The ABR was annualized for each participant using the following formula: ABR = total number of bleeding events/total number of days in the respective period x 365.25. The efficacy period was defined as treatment Day 29 to earlier of end of study date before the dose pause or the last fitusiran administration date before the dose pause + 28 days, whichever comes first for original dose regimen (SAS 1) and the dose re-start Day 169 to the end of study visit for AT-based dose regimen (SAS 2).
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: Full analysis set (FAS) included all participants in SAS.
Measure: Mean (95% Confidence Interval); unit: bleeding events per year
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
bleeding events per year | 3.035 [1.845 to 4.992] | 3.929 [1.622 to 9.520]

9. Secondary Outcome: Annualized Spontaneous Bleeding Rate During the Efficacy Period
Description: A spontaneous bleeding episode was defined as a bleeding event that occurred for no apparent or known reason, particularly into the joints, muscles, and soft tissues. The efficacy period was defined as treatment Day 29 to earlier of end of study date before the dose pause or the last fitusiran administration date before the dose pause + 28 days, whichever comes first for original dose regimen (SAS 1) and the dose re-start Day 169 to the end of study visit for AT-based dose regimen (SAS 2).
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The FAS included all participants in SAS.
Measure: Mean (Standard Deviation); unit: bleeding events per year
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
bleeding events per year | 2.60 (5.96) | 3.96 (11.64)

10. Secondary Outcome: Annualized Joint Bleeding Rate During the Efficacy Period
Description: A joint bleeding episode was defined as an event that is characterized by an unusual sensation in the joint ("aura") in combination with 1) increasing swelling or warmth over the skin over the joint; 2) increasing pain; or 3) progressive loss of range of motion or difficulty in using the limb as compared with baseline. The efficacy period was defined as treatment Day 29 to earlier of end of study date before the dose pause or the last fitusiran administration date before the dose pause + 28 days, whichever comes first for original dose regimen (SAS 1) and the dose re-start Day 169 to the end of study visit for AT-based dose regimen (SAS 2).
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The FAS included all participants in SAS.
Measure: Mean (Standard Deviation); unit: bleeding events per year
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
bleeding events per year | 3.51 (6.97) | 4.78 (11.76)

11. Secondary Outcome: Time Intervals Between Bleeding Events
Description: Bleed-free duration was defined as the time interval between 2 protocol-defined treated bleeding events, excluding events that occurred during the intercurrent periods.
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The FAS included all participants in SAS.
Measure: Median (Full Range); unit: days
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 34 | 18
days | 368.50 [56.0 to 1576.0] | 249.00 [11.0 to 427.0]

12. Secondary Outcome: Annualized Weight-Adjusted Consumption of Coagulation Factor VIII (FVIII) and Coagulation Factor IX (FIX)
Description: Number of coagulation factor injections per bleed was determined. IU= international units, and kg= kilogram.
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The FAS included all participants in SAS. Only participants analyzed for specific factor are reported.
Measure: Mean (Standard Deviation); unit: IU/kg per year
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 11 | 3
IU/kg per year
  FVIII | 63.66 (81.29) | 52.13 (8.50)
  FIXs: number analyzed (Participants) | 5 | 3
  FIXs | 110.26 (93.74) | 108.63 (138.42)

13. Secondary Outcome: Annualized Weight-Adjusted Consumption of Bypassing Agent (BPA) of Recombinant Factor VIIa (rFVIIa)
Description: Number of BPA injections per bleed was determined.
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The FAS included all participants in SAS. Only participants analyzed for specific factor are reported.
Measure: Mean (Standard Deviation); unit: microgram/kg per year
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 5 | 4
microgram/kg per year | 1316.19 (2631.87) | 1431.84 (2369.29)

14. Secondary Outcome: Annualized Weight-Adjusted Consumption of Bypassing Agent (BPA) of Activated Prothrombin Complex Concentrate (aPCC)
Description: Number of BPA injections per bleed was determined.
Time Frame: From Day 29 up to end of the study, maximum of up to 76 months
Population: The FAS included all participants in SAS. Only participants analyzed for this outcome measure are reported.
Measure: Mean (Standard Deviation); unit: units/kg per year
Arm/Group | Original Dose Regimen (SAS 1)
Number analyzed (Participants) | 5
units/kg per year | 381.81 (409.82)

15. Secondary Outcome: Change From Baseline in EuroQoL 5-Dimension 5-level Questionnaire (EQ-5D-5L) Index and Visual Analog Scale (VAS) Scores at Month 24
Description: The EQ-5D-5L is a standardized and disease-generic instrument for use as a measure of quality of life (QoL) outcome. The EQ-5D-5L consists of 2 parts: EQ-5D descriptive system and EQ VAS. The EQ-5D descriptive system included questions for each of following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The VAS recorded participant's self-rated health on a vertical 20-centimeter. VAS scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The EQ-5D-5L questionnaire scores range from 0-100, where 0= worst self-perceived health and 100= best self-perceived health. Positive change from baseline indicates an improvement in QoL. Baseline refers to the last non-missing value on or before the first significant treatment in TDR14767(ALN-AT3SC-001) or LTE14762 study.
Time Frame: Baseline and Month 24
Population: The FAS included all participants in SAS. Only participants analyzed at baseline and Month 24 are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 15 | 3
units on a scale
  Index score | 0.01 (0.14) | 0.09 (0.06)
  VAS score | 4.73 (18.37) | 16.67 (7.64)

16. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life Questionnaire (Haem-A-QoL) Total Score and Physical Health Scores at Month 24
Description: The Haem-A-QoL questionnaire is psychometrically tested QoL assessment instrument for participants with hemophilia and includes 46 items contributing to 10 QoL domains (physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality). Scoring for each item is based on a 5-point Likert scale (1= never, 2= rarely, 3= sometimes, 4= often, and 5= all the time), and the physical health and total transformed scores range from 0 to 100. Higher scores indicated greater impairment. Baseline refers to the last non-missing value on or before the first significant treatment in TDR14767(ALN-AT3SC-001) or LTE14762 study.
Time Frame: Baseline and Month 24
Population: The FAS included all participants in SAS. Only participants analyzed at baseline and Month 24 are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 14 | 3
units on a scale
  Total score | -0.20 (0.47) | 0.02 (0.34)
  Physical health score | -0.14 (0.58) | -0.53 (0.61)

17. Secondary Outcome: Antithrombin Activity Level at the End of Treatment Regimen
Description: The AT activity level was analyzed up to end of treatment regimen. The baseline under the original dose and regimen was the last non-missing assessment before the first significant dose.
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug and had at least 1 blood sample collection post dose to determine plasma AT and thrombin generation (TG) levels.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 16 | 18
percentage | 16.28 (4.53) | 24.76 (7.36)

18. Secondary Outcome: Thrombin Generation at the End of Treatment Regimen
Description: The TG data was analyzed by CoagScope and assay performed using calibrated automated thrombogram method. The baseline under the original dose and regimen was the last non-missing assessment before the first significant dose.
Time Frame: From Day 29 up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months)
Population: The PD analysis set included all participants who received at least 1 dose of study drug and had at least 1 blood sample collection post dose to determine plasma AT and TG levels.
Measure: Mean (Standard Deviation); unit: nanomoles/liter
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
Number analyzed (Participants) | 16 | 18
nanomoles/liter | 71.39 (24.67) | 32.31 (20.05)

19. Secondary Outcome: Maximum Observed Concentration (Cmax) of Fitusiran
Description: Cmax was defined as maximum plasma concentration observed. The non-compartmental Pharmacokinetic (PK) analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1, and Months 12 and 24
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug and have at least 1 blood sample collection post dose to determine plasma concentrations of study drug. Only participants analyzed at each specific time point are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Fitusiran 50 mg: Participants received fitusiran 50 mg QM or Q2M SC injection under original dose regimen (SAS 1) and AT-based dose regimen (SAS 2).
- Fitusiran 80 mg: Participants received fitusiran 80 mg QM SC injection under original dose regimen (SAS 1) and AT-based dose regimen (SAS 2).
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 14 | 17
nanogram per milliliter (ng/mL)
  Day 1 | 86.8 (44.1) | 168 (74.6)
  Month 12: number analyzed (Participants) | 9 | 10
  Month 12 | 75.2 (50.3) | 149 (53.2)
  Month 24: number analyzed (Participants) | 2 | 9
  Month 24 | 62.5 (35.3) | 155 (87.9)

20. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of Fitusiran
Description: tmax was defined as time to reach Cmax. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1, and Months 12 and 24
Population: The PK analysis set included all participants who received at least 1 dose of study drug and have at least 1 blood sample collection post dose to determine plasma concentrations of study drug. Only participants analyzed at each specific time point are reported.
Measure: Median (Full Range); unit: hour
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 14 | 17
hour
  Day 1 | 3.97 [0.50 to 8.08] | 4.00 [2.00 to 8.07]
  Month 12: number analyzed (Participants) | 9 | 10
  Month 12 | 4.02 [2.00 to 8.00] | 6.00 [2.02 to 8.03]
  Month 24: number analyzed (Participants) | 2 | 9
  Month 24 | 4.00 [4.00 to 4.00] | 7.83 [4.05 to 8.00]

21. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to the Real Time (AUClast) of Fitusiran
Description: AUClast was defined as area under the concentration versus time curve from time 0 to the last measurable concentration. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1, and Months 12 and 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 14 | 17
ng*hour/mL
  Day 1 | 1110 (486) | 2130 (769)
  Month 12: number analyzed (Participants) | 9 | 10
  Month 12 | 961 (551) | 2020 (708)
  Month 24: number analyzed (Participants) | 2 | 9
  Month 24 | 935 (550) | 2070 (917)

22. Secondary Outcome: Area Under the Concentration Versus Time Curve Extrapolated to Infinity (AUCinf) of Fitusiran
Description: AUCinf was defined as area under the concentration versus time curve extrapolated to infinity. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1 and Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 4 | 3
ng*h/mL
  Day 1 | 1470 (441) | 2230 (641)
  Month 12: number analyzed (Participants) | 1 | 1
  Month 12 | 356 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | 2860 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

23. Secondary Outcome: Terminal Half-Life (t1/2z) of Fitusiran
Description: t1/2z associated with the terminal slope (λz) determined according to the following equation: t1/2z = 0.693/λz; where, λz is the slope of the regression line of the terminal phase of the plasma concentration versus time curve, in semi-logarithmic scale. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1 and Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 5 | 3
hour
  Day 1 | 5.19 (1.61) | 5.90 (3.83)
  Month 12: number analyzed (Participants) | 1 | 1
  Month 12 | 3.91 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | 4.94 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

24. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Fitusiran
Description: CL/F was defined as apparent clearance of study drug from the body. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1 and Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 4 | 3
liter per hour
  Day 1 | 37.6 (13.6) | 38.8 (12.7)
  Month 12: number analyzed (Participants) | 1 | 1
  Month 12 | 143 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | 28.3 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

25. Secondary Outcome: Apparent Volume of Distribution at the Steady State After Single Extravascular Dose (Vss/F) of Fitusiran
Description: Vss/F was defined as apparent volume of distribution of study drug at steady state concentration. The non-compartmental PK analysis was performed.
Time Frame: Pre-dose and 0.5, 2, 4, 8 and 24 hours post-dose on Day 1 and Month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 4 | 3
liter
  Day 1 | 283 (155) | 390 (348)
  Month 12: number analyzed (Participants) | 1 | 1
  Month 12 | 834 (NA) — Standard deviation could not be determined when only 1 participant was analyzed. | 204 (NA) — Standard deviation could not be determined when only 1 participant was analyzed.

26. Secondary Outcome: Recovery of Fraction of the Dose Excreted in Urine (fe) in 0-24 Hours After Fitusiran Administration
Description: fe was defined as the amount of fitusiran excreted in urine in 0-24 hour. The non-compartmental PK analysis was performed.
Time Frame: Postdose, 0 to 6 hours, 6 to 12 hours, 12 to 24 hours at Month 24
Population: The PK analysis set included all participants who received at least 1 dose of study drug and have at least 1 urine sample collection post dose to determine urine concentrations of study drug. Only those participants with data available at Month 24 are reported.
Measure: Mean (Standard Deviation); unit: percentage of study drug
Arm/Group | Fitusiran 50 mg | Fitusiran 80 mg
Number analyzed (Participants) | 2 | 7
percentage of study drug | 10.7 (4.08) | 12.6 (4.92)

ADVERSE EVENTS:
Time Frame: TEAEs data was collected from first dose of study drug (Day 1) up to end of the study (SAS 1: up to 76 months and SAS 2: up to 40 months).
Description: Analysis was performed on the safety analysis set.
Arm/Group | Original Dose Regimen (SAS 1) | AT-Based Dose Regimen (SAS 2)
All-Cause Mortality (participants affected / at risk) | 1/34 | 0/18
Serious Adverse Events (participants affected / at risk) | 13/34 | 1/18
Other Adverse Events (participants affected / at risk) | 33/34 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Dose Regimen (SAS 1) (N=34) | AT-Based Dose Regimen (SAS 2) (N=18)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (3) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Haemophilic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Dose Regimen (SAS 1) (N=34) | AT-Based Dose Regimen (SAS 2) (N=18)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2 (6) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0)
Erythema Of Eyelid (Eye disorders) | 1 (1) | 0 (0)
Eye Inflammation (Eye disorders) | 0 (0) | 1 (1)
Retinopathy Hypertensive (Eye disorders) | 1 (1) | 0 (0)
Swelling Of Eyelid (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (4) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (5) | 0 (0)
Faeces Pale (Gastrointestinal disorders) | 1 (4) | 0 (0)
Femoral Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Influenza Like Illness (General disorders) | 4 (5) | 0 (0)
Injection Site Atrophy (General disorders) | 1 (1) | 0 (0)
Injection Site Discolouration (General disorders) | 1 (1) | 0 (0)
Injection Site Erythema (General disorders) | 7 (40) | 0 (0)
Injection Site Haematoma (General disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 3 (3) | 0 (0)
Injection Site Swelling (General disorders) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 2 (7) | 0 (0)
Peripheral Swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Swelling Face (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy To Animal (Immune system disorders) | 1 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 2 (2) | 0 (0)
Asymptomatic Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter Infection (Infections and infestations) | 1 (2) | 0 (0)
Herpes Dermatitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Nail Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (13) | 1 (1)
Oral Candidiasis (Infections and infestations) | 2 (4) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (3) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 2 (2) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (8) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (7) | 2 (2)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Paternal Exposure Before Pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Erythema (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Post Procedural Oedema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 10 (15) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 2 (3) | 0 (0)
Fibrin D Dimer Increased (Investigations) | 3 (3) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 3 (3) | 0 (0)
Haematocrit Increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin Increased (Investigations) | 1 (1) | 0 (0)
Prostatic Specific Antigen Increased (Investigations) | 0 (0) | 1 (1)
Protein Urine Present (Investigations) | 1 (1) | 0 (0)
Prothrombin Fragment 1.2 Increased (Investigations) | 1 (1) | 0 (0)
Red Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 5 (9) | 1 (1)
Vitamin D Decreased (Investigations) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (15) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 0 (0)
Haemophilic Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Medial Tibial Stress Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Sacral Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral Cyst (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (21) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitated Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Testicular Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hangnail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pregnancy Of Partner (Social circumstances) | 1 (1) | 0 (0)
Tattoo (Social circumstances) | 1 (1) | 0 (0)
Brachiocephalic Vein Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Collateral Circulation (Vascular disorders) | 1 (1) | 0 (0)
Essential Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Superficial Vein Thrombosis (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT02554773/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02554773/SAP_001.pdf